CLINICAL TRIAL: NCT04523558
Title: Evaluation of the Extended Depth of Focus After Bilateral Implantation of a Hydrophobic IOL With a New Optic Concept Based on a Combination of High Order Aberrations
Brief Title: Evaluation of the Extended Depth of Focus After Bilateral Implantation of Hydrophobic IOLs
Acronym: LuxSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Principal Investigator, Dr. Pavel Stodulka, Chief Eye Surgeon, Gemini Eye Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuxSmart_2020
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cataract Senile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral implantation of LuxSmart hydrophobic IOL (Experimental): Cataract surgery will be carried out using standard phacoemulsification technique with a 2.2 mm incision. Investigators will target a 5.5 mm diameter capsulorhexis to allow the optic to be fully overlapped by the anterior capsular rim.
  The intended target of the post-operative refraction will be emmetropia. The patient will be implanted with LuxSmart hydrophobic IOLs in both eyes and followed up for 6 months
  Interventions: Device: Implantation of LuxSmart hydrophobic IOLs (Bausch + Lomb) in both eyes

INTERVENTIONS:
Device: Implantation of LuxSmart hydrophobic IOLs (Bausch + Lomb) in both eyes — Extended depth of field intraocular lens made form hydrophobic material

SUMMARY:
This will be a prospective observational, ethics committee approved study where patients undergoing routine cataract surgery will have bilateral implantation of the intraocular lens (LuxSmart, Bausch & Lomb). The device under investigation is CE-mark approved and commercially available. The device under investigation and all study products, including the devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

Investigator is accredited and experienced cataract surgeon and researchers who have been involved in similar studies in the past.

The device under investigation LuxSmart (Bausch & Lomb) is a hydrophobic, acrylic copolymer containing UV absorber intraocular lens (IOL). The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

In total 30 patients will be recruited for this first clinical experience and receive bilateral implantation of the LuxSmart. The maximum time between 1st and 2nd eye implantation is 30 days, some patients may receive bilateral implantation on the same day. However there will be a minimum of 1 week between the implantations in the first 10 patients.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity;
* Calculated IOL power is within the range of the study IOLs;
* Male or female adults ages 50 years or older on the day of screening who have cataract(s) in one or both eyes;
* Regular corneal astigmatism ≤1.5D (measured by an automatic keratometry) in one or both eyes;
* Clear intraocular media other than cataract;
* Dilated pupil size large enough to visualize IOL axis markings postoperatively
* Availability, willingness, skills and cognitive awareness enough to comply with the follow-up/study procedures and study visits.
* Subjects able to read, understand and provide written Informed Consent Form on the Ethics Committee approved Informed Consent Form and provide authorization as appropriate for local privacy regulations.

Exclusion Criteria:

* Age of patient <50 years;
* Regular corneal astigmatism >1.5D (measured by an automatic keratometry) in both eyes;
* Irregular astigmatism;
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse;
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema;
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* History or presence of macular edema;
* Instability of keratometry or biometry measurements;
* Advanced or decompensated glaucoma;
* Significant dry eye;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity | 6 months
  Measurement of distance visual acuity is measured with 5 letters modified Snellen charts placed at 6 m distance with corrective glasses for each eye separately

SECONDARY OUTCOMES:
Manifest refraction (sphere, cylinder, axis) | 6 months
  Standard refraction technique
Monocular Uncorrected Distance Visual Acuity (UDVA) | 6 months
  Measurement of distance visual acuity is measured with 5 letter modified snellen charts placed at 6 m distance without corrective glasses for each eye separately
Binocular Uncorrected Distance Visual Acuity (UDVA) | 6 months
  Measurement of distance visual acuity is measured with 5 letter modified snellen charts placed at 6 m distance without corrective glasses for both eyes together
Monocular Corrected Distance Visual Acuity (CDVA) | 6 months
  Measurement of distance visual acuity is measured with 5 letter modified snellen charts placed at 6 m distance with corrective glasses for each eye separately
Binocular Corrected Distance Visual Acuity (CDVA) | 6 months
  Measurement of distance visual acuity is measured with 5 letter modified snellen charts placed at 6 m distance with corrective glasses for both eyes together
Monocular Uncorrected Intermediate Visual Acuity (UIVA) | 6 months
  Measurement performed using ETDRS chart at 66 cm and 80 cm distance for one eye
Binocular Uncorrected Intermediate Visual Acuity (UIVA) | 6 months
  Measurement performed using ETDRS chart at 66 cm and 80 cm distance for both eyes
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) | 6 months
  Measurement performed using ETDRS chart at 66 cm and 80 cm distance for one eye
Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) | 6 months
  Measurement performed using ETDRS chart at 66 cm and 80 cm distance for both eyes
Monocular Defocus Curve | 6 months
  Standard defocus curve with -5.0 to +1.5 D range lenses
Monocular Contrast Sensitivity under photopic and mesopic conditions | 6 months
  Measurement of contrast sensitivity at 2.5 m
Change in the 9-item Catquest short-form questionnaire (Catquest-9SF) score | 6 months
  To assess if difficulties in daily life occur due to impaired sight. This questionnaire is 9-item Rasch-scaled instrument to assess subjective perception of visual impairment after surgery. There are five text response options for the answers scaled from "Yes, very great difficulties" to "No, no difficulties" including answer "Cannot decide". Outcome is a sum score (min: 9, max: 36, lower scores mean a better result)
Overall Spectacle independence | 6 months
  Percent of all patients who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire, or PRSIQ - "a little of the time" or "none of the time".

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, Principal Investigator — Gemini Eye Clinic
Locations (1):
- Gemini Eye Clinic, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: No